CLINICAL TRIAL: NCT00686608
Title: Hypothalamic fMRI Response to Nutrients
Brief Title: Hypothalamic Functional Magnetic Resonance Imaging (fMRI) Response to Nutrients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan Purnell, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: eIRB #938; 791 (Other: Oregon Clinical and Translational Research Institute)
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Glucose; Fructose; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will receive infusions of glucose, fructose, and saline in a randomized order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glucose (Experimental): IV glucose
  Interventions: Dietary Supplement: glucose
- Fructose (Active Comparator)
  Interventions: Dietary Supplement: fructose
- Saline (Placebo Comparator)
  Interventions: Dietary Supplement: saline

INTERVENTIONS:
Dietary Supplement: glucose — 0.3mg/kg of glucose
  Arms: Glucose
Dietary Supplement: fructose — fructose IV bolus
  Arms: Fructose
Dietary Supplement: saline — IV saline
  Arms: Saline

SUMMARY:
The purpose of this study is to identify how certain parts of the brain that control appetite respond to changes in dietary carbohydrate and fat.

DETAILED DESCRIPTION:
To measure fMRI signal change in hypothalamic and brainstem centers associated with control of food intake and energy expenditure in response to IV glucose, fructose, and saline. The fMRI response to these nutrients will then be compared in obese vs. lean subjects. Frequently timed blood samples will be obtained for measurement of nutrients (i.e., glucose) and blood levels of other factors (i.e., insulin, ghrelin, lactate) during these infusion protocols, and to test associations between these levels and the fMRI response.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 year to 45 years of age
* BMI 18 to 25 kg/m2 (25 subjects) and 30 to 40 kg/m2 (25 subjects), matched for age and sex.
* At maximal lifetime weight.
* Weight stable for at least 3 months.

Exclusion Criteria:

* Those with a major medical illness or who require prescription medication, including: cancer, coronary artery disease, hypertension, and diabetes.
* Subjects taking psychiatric or centrally-acting (CNS) medications, or who are diagnosed with a psychiatric or neurological illness, including: depression, anorexia, bulimia, and seizure disorder.
* Subjects who have lost weight as a result of dieting, pharmacological treatment, or bariatric surgery.
* Weight > 350 lbs or girth > 60 inches (the limits of the MR machine)
* Exercise > 30 minutes, 3 times a week.
* Alcohol consumption > 2 drinks / day.
* Weight > 300 lbs (150 kg) (weight limit for MR machine).
* Blood glucose > 100 mg/dL, abnormal creatinine or liver function tests.
* Illicit drug use.
* Pregnancy.
* Extreme dietary habits as determined by a GCRC nutritionist: very high or low dietary carbohydrate, protein, or fat intakes.
* Those with a contraindication to exposure to strong magnetic fields: presence of metal in the body such as body piercing, shrapnel, cardiac pacemakers or aneurysm clips.
* Those with claustrophobia.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2006-10-01 (Actual); Primary Completion 2012-07-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
The primary outcomes of this aim will be the change in fMRI response in the hypothalamus to IV glucose, to IV glucose during intralipid infusion, and to the IV glucose alone, in the lean and obese groups separately. | 0,1,2 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Q. Purnell, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States